CLINICAL TRIAL: NCT02118753
Title: The Effect of Eplerenone on Ischemia Reperfusion Injury in Human Myocardium (EPLICARD Study)
Brief Title: The Effect of EPLerenone on Ischemia Reperfusion Injury in Human myoCARDium
Acronym: EPLICARD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EPLICARD
Record Dates: First submitted 2014-03-14; First posted 2014-04-21 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Ischemia-reperfusion Injury
Keywords: ischemia-reperfusion injury
MeSH Terms: conditions — Reperfusion Injury | interventions — Eplerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ischemic preconditioning (No Intervention): After baseline recordings of contractile function, the investigators will assign 2 trabeculae of each patient to either a stimulus for (1) ischemic preconditioning (IP) or (2) no IP. Subsequently, the trabeculae will be exposed to 90 min of ischemia, followed by 120 minutes of recovery. The investigators will measure the recovery of contractile function in both trabeculae.
  This experiment serves as a positive control, to ensure that our model is still working properly.
- eplerenone (Experimental): In the next patients, a similar ischemia-reperfusion experiment will be performed, but now the 2 trabeculae will be randomized to pretreatment with eplerenone or DMSO. The percentage recovery (compared to baseline) of contractile force of the trabeculae at the end of reperfusion will serve as the primary endpoint.
  Interventions: Drug: Eplerenone

INTERVENTIONS:
Drug: Eplerenone — eplerenone administered ex vivo (to the organ bath in which human atrial tissue is exposed)
  Other Names: Inspra
  Arms: eplerenone

SUMMARY:
In the laboratory, the researchers will investigate whether the drug eplerenone improves contractile function after ischemia and reperfusion in heart tissue.

DETAILED DESCRIPTION:
In animal studies, the mineralocorticoid receptor antagonist eplerenone appears to limit myocardial infarct size. This cardioprotective effect might explain, at least in part, the beneficial effect on mortality of eplerenone in patients with heart failure. Previous animal studies suggest that this cardioprotective effect is mediated by an increased formation of the endogenous nucleoside adenosine.

Our objective is to study for the first time in human myocardial tissue ex vivo wether eplerenone limits ischemia reperfusion injury and whether this is mediated by adenosine receptor stimulation.

From patients undergoing open heart surgery, the right atrial appendage will be harvested by the cardiothoracic surgeon. In the laboratory, two trabeculae will be dissected and suspended in an organ bath. Contraction will be induced by electrical field stimulation. Recovery of contractile force after a period of simulated ischemia and reperfusion will be used as an endpoint of ischemia-reperfusion injury.

The trabeculae of each patient will be randomized to pretreatment with A)ischemic preconditioning (IP) of no IP as a positive control experiment; B)eplerenone or vehicle; C)eplerenone with or without caffeine; and D)aldosterone with and without eplerenone.

ELIGIBILITY:
Inclusion Criteria:

* age>18 years
* willing to sign informed consent
* planned elective surgery with extracorporal circulation

Exclusion Criteria:

* use of theophylline
* use of sulfonylureas
* use of oral antiarrhythmics (not beta blockers)
* use of dipyridamole, use of mineralocorticoid receptor antagonists
* atrial arrhythmias
* right ventricular failure
* known atrial enlargement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-03; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
contractile function after simulated ischemia and reperfusion in response to eplerenone | 210 minutes
  The recovery of contractile function (% of baseline) in human myocardial tissue after simulated ischemia and reperfusion in 2 trabeculae will be compared: 1 of the trabeculae will be exposed to eplerenone, the other to vehicle.
  We will use the experimental set up as described by Speechly-Dick et al. with small modifications to allow simultaneous measurement of 2 trabeculae from 1 patient. The two trabeculae will be dissected and vertically suspended in an organ bath and linked to a force transducer. During electrical field stimulation, we will calculate the developed force (difference between maximal tension during contraction and minimal tension during relaxation), maximal speed of tension development during contraction and maximal speed of tension during relaxation. We will average these parameters for baseline, and during the experiment. Functional recovery will be expressed as a percentage of baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Niels P. Riksen, Dr, Principal Investigator — Radboud University Medical Center; Henri A. van Swieten, Prof dr ir, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Medical Centre, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Background] Riksen NP, Zhou Z, Oyen WJ, Jaspers R, Ramakers BP, Brouwer RM, Boerman OC, Steinmetz N, Smits P, Rongen GA. Caffeine prevents protection in two human models of ischemic preconditioning. J Am Coll Cardiol. 2006 Aug 15;48(4):700-7. doi: 10.1016/j.jacc.2006.04.083. Epub 2006 Jul 24. PMID 16904537
- [Background] Speechly-Dick ME, Grover GJ, Yellon DM. Does ischemic preconditioning in the human involve protein kinase C and the ATP-dependent K+ channel? Studies of contractile function after simulated ischemia in an atrial in vitro model. Circ Res. 1995 Nov;77(5):1030-5. doi: 10.1161/01.res.77.5.1030. PMID 7554138